CLINICAL TRIAL: NCT05661344
Title: Pharmacokinetics, Safety and Tolerability of BI 1015550 Following Oral Administration in Male and Female Participants With Different Degrees of Hepatic Impairment (Child-Pugh Classification A and B) Compared With Matched Male and Female Participants With Normal Hepatic Function (an Open-label, Non-randomised, Single-dose, Parallel, Individual-matched Design Trial)
Brief Title: A Study to Test How BI 1015550 is Taken up in the Blood of People With and Without Liver Problems
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0027; 2022-002811-45 (EudraCT Number)
Record Dates: First submitted 2022-12-15; First posted 2022-12-22 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — BI 1015550

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BI 1015550 mild hepatic impairment (Experimental): Participants with mild hepatic impairment, classified as Child-Pugh A (score 5 to 6 points), administered orally one film-coated tablet of 18 milligram of BI 1015550 with 240 milliliter of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 1015550
- BI 1015550 moderate hepatic impairment (Experimental): Participants with moderate hepatic impairment, classified as Child-Pugh B (score 7 to 9 points), administered orally one film-coated tablet of 18 milligram of BI 1015550 with 240 milliliter of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 1015550
- BI 1015550 normal hepatic function (Experimental): Participants with normal hepatic function administered orally one film-coated tablet of 18 milligram of BI 1015550 with 240 milliliter of water after an overnight fast of at least 10 hours.
  Participants with normal hepatic function were individually matched to participants with mild and/or moderate hepatic impairment. The matching criteria were age (± 10 years), sex and weight (± 15%). One participant with normal hepatic function could match one participant in one or both groups of participants with hepatic impairment.
  Interventions: Drug: BI 1015550

INTERVENTIONS:
Drug: BI 1015550 — BI 1015550
  Other Names: Nerandomilast; JASCAYD®

SUMMARY:
This study is open to adults aged 18 years and older. People without liver problems and people who have mild or moderate liver problems can join the study.

The purpose of this study is to find out how a medicine called BI 1015550 is taken up in the blood of people with and without liver problems. Liver problems may change how a medicine is processed in the body.

Participants are in the study for about 2 weeks. During this time, they visit the study site 6 times. On the second visit, participants stay overnight at the study site for 4 nights. At the visits, doctors take blood samples to measure the levels of BI 1015550 in participants' blood. Then they compare the results between the groups of participants with and without liver problems. The doctors also check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria applicable to all participants

* Male or female participants
* Age 18-79 years (inclusive)
* Body Mass Index (BMI) of 18.5 to 35 kilogram per square meter (kg/m2) (inclusive)
* Signed and dated written informed consent in accordance with Guideline for Guideline for Good Clinical Practice - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Male participants are not required to use contraception
* Women of childbearing potential are allowed to participate provided they use a highly effective contraception from at least 30 days before the administration of trial medication until 7 days after trial completion. Of note, oral hormonal contraceptives are not considered as highly effective in this study due to the potential CYP3A induction by BI 1015550. Methods of contraception considered adequate for female participants of childbearing potential are listed in the protocol.

Inclusion criteria applying only to participants with impaired hepatic function

* Hepatic impairment classified as Child-Pugh A (score 5-6 points) or Child-Pugh B (score 7-9 points)
* further inclusion criteria apply

Inclusion criteria applying only to participants with normal hepatic function

* Individually matched to participants with hepatic impairment according to sex, age, and weight
* further inclusion criteria apply

Exclusion criteria applying to all participants

* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetic(s) (PK) of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (CNS) (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders (including but not limited to major depressive disorder)
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Relevant chronic or acute infections
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin or squamous cell carcinoma in situ of the skin or in situ carcinoma of uterine cervix
* further exclusion criteria apply

Exclusion criteria applying only to participants with hepatic impairment

* A marked prolongation of time from the start of the Q wave to the end of the T wave (QT)/ QT corrected for heart rate (QTc) interval (such as QT Corrected by the Fridericia Formula (QTcF) intervals that are repeatedly greater than 480 milliseconds (ms) in males or repeatedly greater than 500 ms in females) or any other relevant Electrocardiogram (ECG) finding at screening
* further exclusion criteria apply

Exclusion criteria applying only to participants with normal hepatic function

* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR) or ECG) deviating from normal and assessed as clinically relevant by the investigator
* further exclusion criteria apply

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed as a non-randomised, single-dose, open-label, parallel, individual matched design in order to investigate pharmacokinetic(s) of BI 1015550, as well as safety and tolerability of BI 1015550 in male and female participants with mild and moderate hepatic impairment compared to individually matched control participants.
Pre-assignment Details: All participants were screened for eligibility prior to participation in the trial. Participants attended a specialist site which ensured that the participants strictly met all inclusion and none of the exclusion criteria. Participants were not to be entered in the trial if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | BI 1015550 mild hepatic impairment | BI 1015550 moderate hepatic impairment | BI 1015550 normal hepatic function
Started | 8 | 8 | 12
Treated | 8 | 8 | 12
Completed | 8 | 8 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) included all participants who were treated with 1 dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1015550 Mild Hepatic Impairment | BI 1015550 Moderate Hepatic Impairment | BI 1015550 Normal Hepatic Function | Total
Number analyzed (Participants) | 8 | 8 | 12 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (5.5) | 61.0 (7.4) | 64.7 (9.04) | 64.0 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 6 | 14
  Male | 4 | 4 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 8 | 12 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of R-BI 1015550 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of R-BI 1015550 (the pharmacologically active enantiomer, determined using the chiral bioanalytical assay) in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included the effect 'degree of hepatic impairment' as a fixed effect and 'matched pair' as random effect. These quantities were then back-transformed to the original scale.
  The model was fitted separately for the two hepatic impaired groups.
Time Frame: Within the 2 hours before and 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 24, 36, 48, 72, 96, 120 and 144 hours after drug administration.
Population: The pharmacokinetic parameter analysis set (PKS) included all participants in the treated set who provided at least 1 primary or secondary PK endpoint and who were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
  Thus, a participant was to be included in the PKS even if they contributed only 1 of the main PK parameter value to the statistical assessment. Descriptive and model-based analyses of PK parameters were based on the PKS.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomole/liter (h*nmol/L)
Groups:
- BI 1015550 normal hepatic function matched to mild hepatic impairment: Participants with normal hepatic function administered orally one film-coated tablet of 18 milligram of BI 1015550 with 240 milliliter of water after an overnight fast of at least 10 hours.
  Participants with normal hepatic function were individually matched to participants with mild hepatic impairment. The matching criteria were age (± 10 years), sex and weight (± 15%).
- BI 1015550 normal hepatic function matched to moderate hepatic impairment: Participants with normal hepatic function administered orally one film-coated tablet of 18 milligram of BI 1015550 with 240 milliliter of water after an overnight fast of at least 10 hours.
  Participants with normal hepatic function were individually matched to participants with moderate hepatic impairment. The matching criteria were age (± 10 years), sex and weight (± 15%).
Arm/Group | BI 1015550 mild hepatic impairment | BI 1015550 moderate hepatic impairment | BI 1015550 normal hepatic function matched to mild hepatic impairment | BI 1015550 normal hepatic function matched to moderate hepatic impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*nanomole/liter (h*nmol/L) | 2913.55 (NA) — Adjusted geometric standard error = 1.09 | 2837.74 (NA) — Adjusted geometric standard error = 1.16 | 2786.43 (NA) — Adjusted geometric standard error = 1.09 | 2168.11 (NA) — Adjusted geometric standard error = 1.16
Statistical Analysis 1: Comparison: BI 1015550 mild hepatic impairment vs BI 1015550 normal hepatic function matched to mild hepatic impairment; Ratio of adjusted geometric means was calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included the effect 'degree of hepatic impairment' as a fixed effect and 'matched pair' as random effect. These quantities were then back-transformed to the original scale; Test type: Other; Ratio of adjusted geometric means [%] = 104.56, 90% CI 2-sided [91.89 to 118.98] — Ratio [%] = (adjusted geometric mean of mild hepatic impairment / adjusted geometric mean of normal hepatic function matched to mild hepatic impairment)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 13.7
Statistical Analysis 2: Comparison: BI 1015550 moderate hepatic impairment vs BI 1015550 normal hepatic function matched to moderate hepatic impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 130.89, 90% CI 2-sided [89.34 to 191.75] — Ratio [%] = (adjusted geometric mean of moderate hepatic impairment / adjusted geometric mean of normal hepatic function matched to moderate hepatic impairment)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 42.0

2. Primary Outcome: Maximum Measured Concentration of R-BI 1015550 in Plasma (Cmax)
Description: Maximum measured concentration of R-BI 1015550 (the pharmacologically active enantiomer, determined using the chiral bioanalytical assay) in plasma (Cmax) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included the effect 'degree of hepatic impairment' as a fixed effect and 'matched pair' as random effect. These quantities were then back-transformed to the original scale.
  The model was fitted separately for the two hepatic impaired groups.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/liter (nmol/L)
Arm/Group | BI 1015550 mild hepatic impairment | BI 1015550 moderate hepatic impairment | BI 1015550 normal hepatic function matched to mild hepatic impairment | BI 1015550 normal hepatic function matched to moderate hepatic impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
nanomole/liter (nmol/L) | 409.35 (NA) — Adjusted geometric standard error = 1.15 | 277.67 (NA) — Adjusted geometric standard error = 1.19 | 491.48 (NA) — Adjusted geometric standard error = 1.15 | 404.46 (NA) — Adjusted geometric standard error = 1.19
Statistical Analysis 1: Comparison: BI 1015550 mild hepatic impairment vs BI 1015550 normal hepatic function matched to mild hepatic impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 83.29, 90% CI 2-sided [60.47 to 114.71] — Ratio [%] = (adjusted geometric mean of mild hepatic impairment / adjusted geometric mean of normal hepatic function matched to mild hepatic impairment)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 34.8
Statistical Analysis 2: Comparison: BI 1015550 moderate hepatic impairment vs BI 1015550 normal hepatic function matched to moderate hepatic impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 68.65, 90% CI 2-sided [46.48 to 101.41] — Ratio [%] = (adjusted geometric mean of moderate hepatic impairment / adjusted geometric mean of normal hepatic function matched to moderate hepatic impairment)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 43.0

3. Secondary Outcome: Area Under the Concentration-time Curve of R-BI 1015550 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of R-BI 1015550 (the pharmacologically active enantiomer, determined using the chiral bioanalytical assay) in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included the effect 'degree of hepatic impairment' as a fixed effect and 'matched pair' as random effect. These quantities were then back-transformed to the original scale.
  The model was fitted separately for the two hepatic impaired groups.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomole/liter (h*nmol/L)
Arm/Group | BI 1015550 mild hepatic impairment | BI 1015550 moderate hepatic impairment | BI 1015550 normal hepatic function matched to mild hepatic impairment | BI 1015550 normal hepatic function matched to moderate hepatic impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*nanomole/liter (h*nmol/L) | 2964.46 (NA) — Adjusted geometric standard error = 1.09 | 2866.58 (NA) — Adjusted geometric standard error = 1.16 | 2811.48 (NA) — Adjusted geometric standard error = 1.09 | 2186.53 (NA) — Adjusted geometric standard error = 1.16
Statistical Analysis 1: Comparison: BI 1015550 mild hepatic impairment vs BI 1015550 normal hepatic function matched to mild hepatic impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 105.44, 90% CI 2-sided [92.36 to 120.38] — Ratio [%] = (adjusted geometric mean of mild hepatic impairment / adjusted geometric mean of normal hepatic function matched to mild hepatic impairment)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 14.1
Statistical Analysis 2: Comparison: BI 1015550 moderate hepatic impairment vs BI 1015550 normal hepatic function matched to moderate hepatic impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 131.10, 90% CI 2-sided [89.96 to 191.05] — Ratio [%] = (adjusted geometric mean of moderate hepatic impairment / adjusted geometric mean of normal hepatic function matched to moderate hepatic impairment)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 41.4

ADVERSE EVENTS:
Time Frame: From the administration of BI 1015550, until the end of the on-treatment period, up to 7 days. All-cause mortality was recorded from the administration of BI 1015550 until the end of trial, up to 2 weeks.
Description: Treated set (TS) included all participants who were treated with 1 dose of trial drug.
  Adverse events are reported by impairment group according to the Statistical Analysis Plan. The sum of matched controls to the renal impairment groups (16) does not match the number of total participants with normal hepatic function (12), because 4 controls were matched to 1 participant with mild hepatic impairment and to 1 participant with moderate hepatic impairment.
Arm/Group | BI 1015550 normal hepatic function matched to mild hepatic impairment | BI 1015550 mild hepatic impairment | BI 1015550 normal hepatic function matched to moderate hepatic impairment | BI 1015550 moderate hepatic impairment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 2/8 | 1/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1015550 normal hepatic function matched to mild hepatic impairment (N=8) | BI 1015550 mild hepatic impairment (N=8) | BI 1015550 normal hepatic function matched to moderate hepatic impairment (N=8) | BI 1015550 moderate hepatic impairment (N=8)
Headache (Nervous system disorders) | 2 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Catheter site inflammation (General disorders) | 0 | 1 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT05661344/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/44/NCT05661344/SAP_001.pdf